CLINICAL TRIAL: NCT04893837
Title: Non-Invasive Monitoring of Traumatic Brain Injury Progression Using the Infrascanner (MOBI-1)
Acronym: MOBI-1
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); InfraScan, Inc. (Industry)
Responsible Party: Principal Investigator, Jan O. Jansen, Professor and Director, UAB Center for Injury Science, University of Alabama at Birmingham
Other Study IDs: IRB-300007257; 20-15-TBI-008 (Other Grant/Funding Number: MTEC)
Record Dates: First submitted 2021-05-14; First posted 2021-05-20 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Brain Injuries, Traumatic
Keywords: traumatic brain injury, TBI, intracranial hematoma, ICH
MeSH Terms: conditions — Brain Injuries, Traumatic; Hepatitis, Infectious Canine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Standard care plus infrascans: All participants will receive regular clinical neurological assessments as ordered by the clinical care team. In addition, a research team member will perform an infrascan. This process will be repeated hourly at the same timepoint as the clinical neurological assessments. If a patient's neurological status deteriorates at any time point, and the medical team orders an early (unplanned) CT scan, the neurological data collection will cease once the patient is sent to CT.
  Infrascan results will not be shared with the clinical care team, and will not guide the participants' care in any way.
  Interventions: Device: Standard care plus infrascans

INTERVENTIONS:
Device: Standard care plus infrascans — Hourly infrascans to detect expanding intracranial hematomas

SUMMARY:
MOBI-1 is a multicenter clinical trial that will evaluate the use of the Infrascanner for the monitoring of traumatic intracranial hematomas.

DETAILED DESCRIPTION:
MOBI-1 is a single-arm, multi-center derivation / validation study that will evaluate the use of the Infrascanner for monitoring traumatic intracranial hematomas. All patients will receive standard care plus hourly infrascanner assessments. This study will test the hypotheses that:

1. The Infrascanner has sufficient diagnostic performance to detect the expansion of intracranial hematomas
2. Patients who have expanding intracranial hematomas will be identified faster when monitored with hourly infrascanner assessments compared to standard care alone
3. Clinical / research staff will be able to attain all data points and relay the assessments to the medical team.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15 or older
2. Admission CT Scan shows intracranial hemorrhage
3. Glasgow Coma Scale less than 15
4. Neurosurgery service determines initial care is nonoperative
5. Admitted for observation for TBI, to either step-down unit or intensive care unit

Exclusion Criteria:

1. Inability to provide informed consent or lack of a legally authorized representative (LAR)
2. Admitted and observed for >2 hours prior to screening (i.e., has already received second neurological check)
3. Other injuries deemed non-survivable
4. Diagnosed with hemorrhagic shock or receives a large volume transfusion (>3 units of any blood product within any 1 hour)
5. Planned surgical interventions/ procedures during study period (before the second CT scan)
6. Known prisoner

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll up to 440 patients over 14 months, at 10 trauma centers. Currently, there are no high quality published datasets or literature to document the mean or variability in time to the detection of hematoma expansion that could be used for meaningful sample size projections. Therefore, this study has been designed to provide reasonable estimates of the future study outcomes.
Sampling Method: Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of the infrascanner | Month 24
  Number of participants whose Infrascan results were accurate

SECONDARY OUTCOMES:
Time to detection of an enlarging hematoma | 0-12 hours
  Difference in time to detection of hematoma enlargement between Infrascan and second CT across the cohort

CONTACTS AND LOCATIONS:
Overall Officials: Jan O Jansen, MBBS, PhD, Principal Investigator — University of Alabama at Birmingham, Center for Injury Science
Locations (2):
- United States (2):
  - UAB Hospital, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: Yes
This data will be uploaded to the Federal Interagency Traumatic Brain Injury Research (FITBIR) informatics system, as a requirement of the funding agency. Only de-identified data will be shared.
Time Frame: Data will be uploaded to FITBIR annually.
Access Criteria: Access is through the FITBIR system, per their requirements.
URL: https://fitbir.nih.gov/